CLINICAL TRIAL: NCT02473120
Title: Determination of ESR1 Mutations by Digital PCR During Aromatase Inhibitor Treatment in Metastatic Breast Cancer
Brief Title: Study of ESR1 Mutations in Metastatic Breast Cancer
Acronym: FMER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHB 15.01
Record Dates: First submitted 2015-06-08; First posted 2015-06-16 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Metastatic Breast Cancer
Keywords: metastatic; ESR1; aromatase inhibitor; breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Determination of ESR1 mutations (Experimental): Blood sample will be collected every 3 months during two years to determine ESR1 mutations
  Interventions: Biological: Determination of ESR1 mutations

INTERVENTIONS:
Biological: Determination of ESR1 mutations — Blood sample prelevement. Plasma issued from patient with metastatic breast cancer will be analysed at progression by Digital PCR to detect ESR1 mutations

SUMMARY:
The purpose of the study is to determine the frequency ESR1 mutations by Digital PCR in patient with metastatic breast cancer.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer in woman. Aromatase inhibitors have demonstrated a real efficacy however a resistance to treatment exists.

ESR1 mutations appear like involved in the mechanism of resistance to aromatase inhibitors treatment.

The purpose of the study is to determine the frequency ESR1 mutations by Digital PCR in patient with metastatic breast cancer.

The significance of the Digital PCR technique will be determined first in plasma issued from healthy volunteers.

At the initiation of aromatase inhibitors treatment patient with metastatic breast cancer will be included in the study. During their follow-up visit every 3 months), their status towards their disease will be collected and a plasma will be collected too.

When the patient progress clinically or radiologically the plasma concomitant to this progression will be analysed by Digital PCR to detect ESR1 mutations.

The patient will be followed during 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Woman aged superior to 18 years old
* Inform consent signed
* Metastatic breast cancer or loco-regionnaly advanced breast cancer
* Inoperable
* With an indication to treat with aromatase inhibitor
* Treatment with aromatase inhibitors innitiated at the inclusion or at least 6 months before inclusion with a stable disease
* Without precedent treatment or with treatment by chemotherapy/tamoxifen/faslodex or aromatase inhibitors in a adjuvant treatment and with a time frame of 2 years between last treatment with aromatase inhibitors and metastatic evolution
* Treatment by aromatase inhibitors alone or in combination with a targeted therapy (trastuzumab +/- pertuzumab, bevacizumab, everolimus)

Exclusion Criteria:

* No inform consent signed
* Patient under guardianship, curatorship
* Psychosocial disorder
* No affiliated or beneficiary of a social benefit system

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Frequency of ESR1 mutations | up to 24 months
  Determination of the frequency of ESR1 mutation in patient who have a clinical and/or a radiological progression disease

SECONDARY OUTCOMES:
Frequency of progression without ESR1 mutations | up to 24 months
  Determination of frequency of patient with a progression disease and without any ESR1 mutations
Time between introduction of aromatase inhibitor and detection of ESR1 mutations | up to 24 months
  Time between introduction of aromatase inhibitor and detection of ESR1 mutations by digital PCR

CONTACTS AND LOCATIONS:
Overall Officials: Anne Perdrix, MD, Principal Investigator — Centre Henri Becquerel
Locations (1):
- Centre Henri Becquerel, Rouen, France

REFERENCES:
- [Derived] Clatot F, Perdrix A, Beaussire L, Lequesne J, Levy C, Emile G, Bubenheim M, Lacaille S, Calbrix C, Augusto L, Guillemet C, Alexandru C, Fontanilles M, Sefrioui D, Burel L, Guenot S, Richard D, Sarafan-Vasseur N, Di Fiore F. Risk of early progression according to circulating ESR1 mutation, CA-15.3 and cfDNA increases under first-line anti-aromatase treatment in metastatic breast cancer. Breast Cancer Res. 2020 May 28;22(1):56. doi: 10.1186/s13058-020-01290-x. PMID 32466779